CLINICAL TRIAL: NCT04847778
Title: Randomized Clinical Trial to Assess the Efficacy of the System Insulclock® 360 for Insulin Treatment Management in Type 1 Diabetes Patients With Insufficient Glycemic Control
Brief Title: Assess the Impact of Insulclock on Glycemic Variability and Treatment Compliance in Uncontrolled DM1 Patients
Acronym: Segoclock2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital General de Segovia (Other)
Collaborators: Insulcloud S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: INSULCLOCK2018
Record Dates: First submitted 2021-03-24; First posted 2021-04-19 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Type 1 Diabetes Mellitus; Insulin Pen; Glycosylated Hemoglobin; Time in Range; Adherence; Continuous Glucose Monitoring; Insulclock; Basal glycaemia; Preprandial glycaemia; Endocrine System Diseases; Insulin-dependent; Glucose Metabolism Disorders
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Endocrine System Diseases; Glucose Metabolism Disorders

STUDY DESIGN:
Intervention Model Description: All participants will start the study using Insulclock, device and app on Masked Mode. At the week 4 patients will be randomized (1:1) to the Active Insulclock group or the Masked Insulclock group. Patients randomized in the Insulclock Active Group will receive detailed instructions on using the Insulclock device and Insulclock 360 mobile application and will be instructed and motivated for full use of all system functions (alarms, messages to the caregivers and investigation team). Patients randomized in the Insulclock Masked Group will be instructed on the correct installation and use of the Insulclock system for recording insulin bolus information but they will not receive any other information and will not have access to the Insulclock 360 application from the Internet and will keep administering insulin treatment as before. A healthcare professional will apply a FreeStyle Libre sensor to the upper arm in all the participants who do not use a CGM.
Who Masked: Participant
Masking Description: * Patients will be instructed on the correct installation and use of the Insulclock 360 system for recording insulin bolus information.
  * Patients do not receive any other information and will not have access to the Insulclock 360 application from the Internet.
  * They will keep administering insulin treatment as before.
  * Randomization is blind to the recruiting investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Masked arm (Active Comparator): * Participants will be instructed on the correct installation and use of the Insulclock device and app on masked mode for recording insulin bolus information.
  * Participants do not receive any other information and will not have access to the Insulclock 360 application from the Internet.
  * Participants will keep administering insulin treatment as usual.
  Interventions: Device: Use of Insulclock system, both Insulclock device and Insulclock app on masked mode.
- Active arm (Active Comparator): * Participants will receive detailed instructions on using the Insuclock 360 app and Insulclock device
  * Participants will be instructed and motivated for full use of all system functions: alarms, messages to the caregivers and investigation team.
  Interventions: Device: Use of Insulclock system, both Insulclock device and Insulclock 360 app.; Device: Use of Insulclock system, both Insulclock device and Insulclock app on masked mode.

INTERVENTIONS:
Device: Use of Insulclock system, both Insulclock device and Insulclock 360 app. — Visit 5, during week 4.
  Randomization will be applied:
  Active group will use all functionalities of Insulclock 360. They will have reminders, all their information and statistics at the disposition of the patient and healthcare providers, they have the assistance if desired of an ally or caregiver, a bolus calculator and the rest of functionalities described in the protocol.
  Arms: Active arm
Device: Use of Insulclock system, both Insulclock device and Insulclock app on masked mode. — Visit 5, during week 4.
  Randomization will be applied:
  Masked group will remain with the masked system, without functionalities.

SUMMARY:
Insulclock® is a small electronic device developed to facilitate the optimal administration of insulin. This device works as an add-on module of commercially available insulin pens and monitors the date, time and dose of injections, the type of insulin injected, the duration of injections and insulin temperature. The Insulclock 360 app allows automatic data logging, report generation and reminder setting, among other functions. In this study, we pretend to show the clinical impact of Insulclock system, both device and mobile application, on glycemic indices, treatment compliance, and quality of life in patients with persistent poorly controlled T1DM.

Material and methods: Randomized open-label multicenter controlled trial to evaluate glycemic control, the number of missed and delayed insulin doses, and quality of life after seven weeks of Insulclock 360 use in participants with uncontrolled DM1. We will also compare these results between patients with or without receiving system reminders and alerts.

This study aims to assess the effect of Insulclock on glycemic control, treatment adherence, and quality of life. As a secondary objective, we will compare the study outcomes between participants in the Active and Masked Insulclock groups (i.e., with or without receiving alerts and reminders and accessing the app).

To assess glycemic control, we will measure HbA1C and glycemic indices. Glycemic variability indices will be monitored with the FreeStyle Libre™ and included glucose coefficient of variation (CV), standard deviation (SD), time in range (TIR), time above range (TAR), and time below range (TBR). Mean glucose levels will be obtained from 48-h time intervals with the FreeStyle Libre.

A late meal bolus (mistimed) will be considered when Insulclock detects the injection at least 30 minutes after the CGM rise. To identify meal glucose excursions, we will use the Glucose Rate Increase Detector (GRID) algorithm, which estimates the rate of change (ROC) of glucose from CGM data.

Participants will complete the ITSQ and the DTSQ, which are validated questionnaires to assess the diabetes treatment satisfaction.

DETAILED DESCRIPTION:
Study design:

This multicentric randomized open-label study will be conducted at the Hospital General de Segovia (Segovia, Spain), Hospital de Cruces (Bilbao, Spain), Hospital Arquitecto Marcide (Ferrol, A Coruña, Spain) and Hospital Central de Asturias (Oviedo, Spain) after classification by the Spanish Agency for Medicines and Health Products (AEMPS) and ethical approval by the Ethics Review Committee of each research center. The study will be conducted in compliance with the ethical principles of the Declaration of Helsinki. Each participant will provide written informed consent before being included in the study.

The study is scheduled across seven visits. At Visit 1 (Screening, Week -1), demographic and clinical information will be collected, and concomitant medications will be registered. All potential study patients will be screened for eligibility after signing the informed consent form (ICF) and will be assigned with a patient identification number. Laboratory evaluations (HbA1c, serum chemistry) must be available within the last 2 months. An identification number will be assigned to each participant At Visit 2 (Run-in, week 0), participants will receive information on the use of the Insulclock device and app on masked mode (excluding the use of Insulclock 360 app information and alarms). If the participant does not use a CGM: a healthcare professional applies the FreeStyle Libre sensor to the back of the upper arm and activates it. If the participant already uses a CGM system, the patient will be encouraged to use sensors during this period.

At Visit 3 (First Visit CGM 1, week 1) and Visit 4 (Follow-up, week 3), participants will be encouraged to use the system At Visit 5 (Visit Starting CGM 2 and Randomization, week 4) participants will be randomized (1:1) to the Active Insulclock group or the Masked Insulclock group. Participants randomized in the Insulclock Active Group will receive detailed instructions on using the Insulclock device and Insulclock 360 mobile application and will be instructed and motivated for full use of all system functions (alarms, messages to the caregivers and investigation team). Participants randomized in the Insulclock Masked Group will be instructed on the correct installation and use of the Insulclock system for recording insulin bolus information but they will not receive any other information and will not have access to the Insulclock 360 application from the Internet and will keep administering insulin treatment as before. A healthcare professional will apply a FreeStyle Libre sensor to the upper arm in all the participants who do not use a CGM and will be encouraged to wear the sensor for 2 weeks. Participants who already use a CGM system will be encouraged to use sensors during this period.

At Visit 6 (Final Visit CGM 2 and Randomization, week 6). Participants will receive a reminder on the use of Insulclock according to the corresponding group.

At Visit 7 (Final Visit, week 7) the mobile application diaries will be collected and reviewed. Participants will receive to fill in the Insulin Treatment Satisfaction Questionnaire (ITSQ) and the Diabetes Treatment Questionnaire (DTSQ).

Study population Investigators will include 80 participants aged 18-80 years with uncontrolled T1DM who provide written informed consent. Persistent uncontrolled T1DM was defined as HbA1C levels ≥6.5% for at least 1 year, and/or variations ≥1% in HbA1C within the previous 2 years and attending regular (more than 2 per year) follow-up visits at the Endocrinology department. Investigators will exclude pregnant or breastfeeding women, individuals with a history of or current alcohol or drug abuse, acute infection, cognitive decline or dementia, or any illness or condition that could interfere with the trial.

Study devices:

Insulclock is a small electronic device that works as an add-on module of insulin pens. This device can record the dose and time of insulin injected, register temperature changes of insulin pens, record the duration of an injection, and the specific insulin pen used. In the present study, participants self-administer insulin with pens coupled to Insulclock and according to routine clinical practice. By means of acoustic and visual alarms, participants receive information for a correct injection technique (an alert if the injection time was <6 seconds) or to prevent stacking insulin (an alert if a previous injection was done within the 2 previous hours).

The Insulclock device is synchronized with the Insulclock 360 app for the automatic logging of patient data. The Insulclock 360 app also has a reminder function to promote the timely administration of insulin doses. Users can also receive customized tips on DM management with the "my tutors" tool and obtain information on DM topics. Insulclock 360 app is compatible with Apple and Android operating systems.

In the Active group, participants will receive acoustic and visual alarms, device-related information and will have access to the Insulclock 360 app. In the Masked group, participants know the dose, time and duration of injections, but these participants will not receive any reminder and will be masked to the Insulclock 360 app.

Participants will use the Freestyle Libre (Abbott Diabetes Care, Witney, Oxon, UK) for the continuous monitoring of glucose levels. This flash continuous monitoring system is to be worn on the upper arm and does not require capillary glucose concentrations for calibration. The sensor automatically records glucose data every 15 minutes for 14 days.

Statistical Analysis The proposed statistical analysis methods constitute a synthesis of the methods to be used in this study to apply them to the data collected and respond to the general objective and the specific objectives.

Data from all participants included in the study, who meet the selection criteria, will be analyzed. Data in absentia will not be charged and will be considered as lost.

A general description of the variables included in the study will be made. The absolute and relative frequency distributions of the qualitative variables will be presented by investigators, as well as the measures of central tendency and dispersion (mean, standard deviation, median, minimum and maximum) of the quantitative variables. The confidence intervals will be presented at 95% for the main quantitative outcome variables associated with the main objective and the main secondary variables.

The data corresponding to the variables included in the main objective will be descriptively analyzed.

Investigators will use the SPSS software Version 17.0. to perform the analysis. The hypothesis tests that are carried out will be in all bilateral cases and with a significance level of 0.05. For variables that do not fit the normal distribution(or parametric), the Mann Whitney hypothesis tests will be used (for unpaired data). The chi-square test (or Fischer's exact test when appropriate) will be used for the analysis of contingency tables as well as for the comparison of proportions and/or frequency distributions.

ELIGIBILITY:
Inclusion Criteria:

1. age range: 14 to 80 years
2. DM1 diagnosed
3. Patients with type 1 diabetes and poor glycemic control, defined as:

   * HbA1c ≥ 6.5% during more than a year
   * and/or extreme variations (more than 1% of change in HbA1c in the last 2 years)
   * and regular visits to the Endocrinology Unit / Diabetes Unit (more than four each year).
4. Signed informed consent form
5. Ability of the subjects to use the system and fill the included questionnaires
6. Ability and willingness of following and be compatible with the protocol of the clinical trial

Exclusion Criteria:

1. Rejection or inability to give the informed consent to participate in the trial.
2. Pregnancy or lactation
3. Addiction or abuse of alcohol, or history of drug abuse in the last years
4. Dementia diagnosis
5. Acute infection
6. Any illness or condition that, according to investigator, could interfere with the trial

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Change in "Time In Range" (TIR) | Baseline, 7 weeks
  TIR, is the percentage of time that a person spends with their blood glucose levels in a target range. The range will vary depending on the person, but general guidelines suggest starting with a range of 70 to 180 mg/dl. Glucose levels are obtained from Continuous Glucose Monitor (CGM) and investigators compare the results obtained within the first 4 weeks of the study with the values of the next 3 weeks of the study.
Number of daily insulin injections irregularities | Week 0 through week 7
  The number of insulin injections irregularities (omission, mistiming and dosing) will be registered in the Insulclock pen cap device and will be transferred to the Insulclock mobile application in real time to monitor treatment adherence.The moment of the insulin injection will be compared with the moment of food intake analyzing the glycemic excursion. Investigators will determine if the insulin was injected with ahead of time enough, so that catalog the injection as on time, mistiming or omission.

SECONDARY OUTCOMES:
Change in Mean glucose | Baseline, 7 weeks
  Data are collected from the CGM of participants included in the active group, comparing mean glucose levels when patients were in the active group with the mean glucose levels obtained when these participants were included in the masked group.
Change in Diabetes Treatment Satisfaction Questionnaire (DTSQc-change) Score. | Baseline, 7 weeks
  The amplitude of the score on the DTSQc gives the degree of change in satisfaction while the direction (positive or negative) will provide guidance on the preference of one device over the other. DTSQc contains eight items scored on 7-point scales; scores range from +6 = much more satisfied now to 0 = much less satisfied now, with 3 (midpoint), representing no change.
Change in Insulin Treatment Satisfaction Questionnaire (ITSQ-change) Score. | Baseline, 7 weeks
  The ITSQ assesses the perceptions of patients on insulin treatment and their current treatment with insulin and how this affects their daily life.
  ITSQ includes 7 domains: leisure activities, psychological barriers, handling, diabetes control, dependence, weight control, sleep. And 22 items scored on 7-point scales; scores range from +6 = much more satisfied now to 0 = much less satisfied now, with 3 (midpoint), representing no change.

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Gomez Peralta, Physician, Principal Investigator — Hospital General de Segovia, Segovia, Spain
Locations (4):
- Spain (4):
  - Endocrinology and Nutrition Unit, Arquitecto Marcide Hospital, Ferrol, A Coruña
  - Endocrinology and Nutrition Service, Hospital de Cruces., Bilbao
  - Endocrinology and Nutrition Service, Hospital Central de Asturias, Oviedo
  - Endocrinology and Nutrition Unit /Diabetes Unit, Hospital General de Segovia, Segovia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Soriguer F, Goday A, Bosch-Comas A, Bordiu E, Calle-Pascual A, Carmena R, Casamitjana R, Castano L, Castell C, Catala M, Delgado E, Franch J, Gaztambide S, Girbes J, Gomis R, Gutierrez G, Lopez-Alba A, Martinez-Larrad MT, Menendez E, Mora-Peces I, Ortega E, Pascual-Manich G, Rojo-Martinez G, Serrano-Rios M, Valdes S, Vazquez JA, Vendrell J. Prevalence of diabetes mellitus and impaired glucose regulation in Spain: the Di@bet.es Study. Diabetologia. 2012 Jan;55(1):88-93. doi: 10.1007/s00125-011-2336-9. Epub 2011 Oct 11. PMID 21987347
- [Background] American Diabetes Association. 7. Approaches to Glycemic Treatment. Diabetes Care. 2016 Jan;39 Suppl 1:S52-9. doi: 10.2337/dc16-S010. No abstract available. PMID 26696682
- [Background] Borschuk AP, Everhart RS. Health disparities among youth with type 1 diabetes: A systematic review of the current literature. Fam Syst Health. 2015 Sep;33(3):297-313. doi: 10.1037/fsh0000134. Epub 2015 May 18. PMID 25984737
- [Background] Martyn-Nemeth P, Schwarz Farabi S, Mihailescu D, Nemeth J, Quinn L. Fear of hypoglycemia in adults with type 1 diabetes: impact of therapeutic advances and strategies for prevention - a review. J Diabetes Complications. 2016 Jan-Feb;30(1):167-77. doi: 10.1016/j.jdiacomp.2015.09.003. Epub 2015 Sep 7. PMID 26439754
- [Background] Stolpe S, Kroes MA, Webb N, Wisniewski T. A Systematic Review of Insulin Adherence Measures in Patients with Diabetes. J Manag Care Spec Pharm. 2016 Nov;22(11):1224-1246. doi: 10.18553/jmcp.2016.22.11.1224. PMID 27783551
- [Background] Peyrot M, Rubin RR, Kruger DF, Travis LB. Correlates of insulin injection omission. Diabetes Care. 2010 Feb;33(2):240-5. doi: 10.2337/dc09-1348. PMID 20103556
- [Background] Celik S, Cosansu G, Erdogan S, Kahraman A, Isik S, Bayrak G, Bektas B, Olgun N. Using mobile phone text messages to improve insulin injection technique and glycaemic control in patients with diabetes mellitus: a multi-centre study in Turkey. J Clin Nurs. 2015 Jun;24(11-12):1525-33. doi: 10.1111/jocn.12731. Epub 2014 Nov 25. PMID 25422134
- [Background] Arsand E, Muzny M, Bradway M, Muzik J, Hartvigsen G. Performance of the first combined smartwatch and smartphone diabetes diary application study. J Diabetes Sci Technol. 2015 May;9(3):556-63. doi: 10.1177/1932296814567708. Epub 2015 Jan 14. PMID 25591859
- [Background] Klausmann G, Hramiak I, Qvist M, Mikkelsen KH, Guo X. Evaluation of preference for a novel durable insulin pen with memory function among patients with diabetes and health care professionals. Patient Prefer Adherence. 2013 Apr 5;7:285-92. doi: 10.2147/PPA.S41929. Print 2013. PMID 23630416
- [Background] Guo X, Sommavilla B, Vanterpool G, Qvist M, Bethien M, Lilleore SK. Evaluation of a new durable insulin pen with memory function among people with diabetes and healthcare professionals. Expert Opin Drug Deliv. 2012 Apr;9(4):355-6. doi: 10.1517/17425247.2012.671808. PMID 22432521
- [Background] Danne T, Forst T, Deinhard J, Rose L, Moennig E, Haupt A. No effect of insulin pen with memory function on glycemic control in a patient cohort with poorly controlled type 1 diabetes: a randomized open-label study. J Diabetes Sci Technol. 2012 Nov 1;6(6):1392-7. doi: 10.1177/193229681200600619. PMID 23294785
- [Background] Burdick J, Chase HP, Slover RH, Knievel K, Scrimgeour L, Maniatis AK, Klingensmith GJ. Missed insulin meal boluses and elevated hemoglobin A1c levels in children receiving insulin pump therapy. Pediatrics. 2004 Mar;113(3 Pt 1):e221-4. doi: 10.1542/peds.113.3.e221. PMID 14993580
- [Background] Diabetes Control and Complications Trial Research Group; Nathan DM, Genuth S, Lachin J, Cleary P, Crofford O, Davis M, Rand L, Siebert C. The effect of intensive treatment of diabetes on the development and progression of long-term complications in insulin-dependent diabetes mellitus. N Engl J Med. 1993 Sep 30;329(14):977-86. doi: 10.1056/NEJM199309303291401. PMID 8366922
- [Background] Phan TL, Hossain J, Lawless S, Werk LN. Quarterly visits with glycated hemoglobin monitoring: the sweet spot for glycemic control in youth with type 1 diabetes. Diabetes Care. 2014 Feb;37(2):341-5. doi: 10.2337/dc13-0980. Epub 2013 Sep 23. PMID 24062334
- [Background] Luo M, Tan KHX, Tan CS, Lim WY, Tai ES, Venkataraman K. Longitudinal trends in HbA1c patterns and association with outcomes: A systematic review. Diabetes Metab Res Rev. 2018 Sep;34(6):e3015. doi: 10.1002/dmrr.3015. Epub 2018 May 22. PMID 29663623
- [Background] Gomez-Peralta F, Abreu C, Gomez-Rodriguez S, Ruiz L. Insulclock: A Novel Insulin Delivery Optimization and Tracking System. Diabetes Technol Ther. 2019 Apr;21(4):209-214. doi: 10.1089/dia.2018.0361. Epub 2019 Mar 21. PMID 30896261
- [Background] Gomez-Peralta F, Abreu C, Gomez-Rodriguez S, Cruz-Bravo M, Maria-Sanchez C, Poza G, Ruiz-Valdepenas L. Efficacy of Insulclock in Patients with Poorly Controlled Type 1 Diabetes Mellitus: A Pilot, Randomized Clinical Trial. Diabetes Technol Ther. 2020 Sep;22(9):686-690. doi: 10.1089/dia.2019.0427. Epub 2020 Mar 5. PMID 32069067
- [Background] Ruiz-Ramos M, Escolar-Pujolar A, Mayoral-Sanchez E, Corral-San Laureano F, Fernandez-Fernandez I. [Diabetes mellitus in Spain: death rates, prevalence, impact, costs and inequalities]. Gac Sanit. 2006 Mar;20 Suppl 1:15-24. doi: 10.1157/13086022. Spanish. PMID 16539961
- See also: Homepage of the Insuclock device and Insulclock 360 app — https://www.insulcloud.com/

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2021-01-09): https://cdn.clinicaltrials.gov/large-docs/78/NCT04847778/Prot_ICF_000.pdf